CLINICAL TRIAL: NCT00679653
Title: Blood Pressure and Weight Trajectory on a Dual Antihypertensive Combination Plus Sibutramine Versus Placebo in Obese Hypertensives
Acronym: HOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Prof. Dr. Med J. Scholze, Director of Charite Medical OPD
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KD200010
Record Dates: First submitted 2008-03-26; First posted 2008-05-19 (Estimated); Last update posted 2008-05-19 (Estimated); Status verified 2008-05

CONDITIONS: Obesity; Hypertension
MeSH Terms: conditions — Obesity; Hypertension | interventions — sibutramine; Verapamil; trandolapril; Felodipine; Ramipril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): verapamil/trandolapril
  Interventions: Drug: sibutramine; Drug: verapamil/trandolapril
- 2 (Active Comparator): metoprolol/HCT
  Interventions: Drug: sibutramine; Drug: metoprolol/HCT
- 3 (Active Comparator): felodipine/ramipril
  Interventions: Drug: sibutramine; Drug: felodipine/ramipril

INTERVENTIONS:
Drug: sibutramine — 8-wks, sibutramine, 10 mg, capsules, once daily
  Other Names: ABT-991; Meridia; Reductil
Drug: sibutramine — 8-wks, sibutramine, 15 mg, capsules, once daily
  Other Names: ABT-991; Meridia; Reductil
Drug: verapamil/trandolapril — 2 wk Run-in phase, antihypertensive therapy only
  Arms: 1
Drug: metoprolol/HCT — 2 wk Run-in phase, antihypertensive therapy only
  Arms: 2
Drug: felodipine/ramipril — 2 wk Run-in phase, antihypertensive therapy only
  Arms: 3

SUMMARY:
To study the effect of sibutramine treatment on weight reduction and blood pressure improvement in three groups with antihypertensive therapy whose blood pressure was not adequately controlled with antihypertensive combination treatment.

ELIGIBILITY:
Inclusion Criteria:

* Treated essential hypertension.
* Obesity: BMI 27-35 kg/m2

Exclusion Criteria:

* Secondary hypertension.
* Stage 3 hypertension.
* Secondary obesity; BMI > 35kg/m2.
* CAD; MI within past 6 months; NYHA stage 3 or 4 heart failure; tachyarrhythmia/atrial fibrillation; myocarditis.
* Kidney failure.
* Liver failure.
* Hyperthyroidism.
* Unstable DM.
* Carcinoma.
* Severe chronic infectious disease.
* Alcohol or drug abuse.
* Pregnancy.
* Epilepsy.
* Psychosis or treatment with antidepressants or major tranquilizers

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2002-02; Primary Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | Duration of Study
Diastolic Blood Pressure | Duration of Study